CLINICAL TRIAL: NCT00549198
Title: Study of Once-Daily Abacavir/Lamivudine Versus Tenofovir/Emtricitabine, Administered With Efavirenz in Antiretroviral-Naive, HIV-1 Infected Adult Subjects
Brief Title: KIVEXA Vs TRUVADA, Both Administered With Efavirenz, In ART-Naive Subjects
Acronym: ASSERT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNA109586
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: tenofovir; HIV; efavirenz; naive; lamivudine; abacavir; emtricitabine; renal
MeSH Terms: conditions — Infections; HIV Infections | interventions — abacavir; Lamivudine; efavirenz; Tenofovir; Emtricitabine

ARMS (2):
- ABC/3TC + EFV (Experimental)
  Interventions: Drug: Abacavir/lamivudine and efavirenz
- TDF/FTC + EFV (Active Comparator)
  Interventions: Drug: Tenofovir/Emtricitabine and efavirenz

INTERVENTIONS:
Drug: Abacavir/lamivudine and efavirenz
  Arms: ABC/3TC + EFV
Drug: Tenofovir/Emtricitabine and efavirenz
  Arms: TDF/FTC + EFV

SUMMARY:
Recently, the fixed-dose combinations (FDC) KIVEXA™ (abacavir/lamivudine) and TRUVADA (tenofovir disoproxil fumarate/emtricitabine) have facilitated the usage of once-daily regimens. However data from head-to-head randomized trials comparing these two FDCs as part of an initial regimen are not available at present. The long-term toxicity profiles of these regimens are of particular importance, as treatment of HIV is currently life-long and therefore, minimizing long-term toxicity and maximizing adherence and duration of regimen maintenance are critical therapy objectives.

The primary endpoint is estimated glomerular filtration rate (GFR), as measured by the modified diet in renal disease (MDRD) equation, a validated estimate of renal function.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject is antiretroviral-naïve (defined as having no previous therapy with any NNRTI and 14 days of prior therapy with any other antiretroviral).
* Subject has plasma HIV-1 RNA 1,000 copies/mL at screening. This test may be repeated once within the 45-day screening window.
* Subject is willing and able to understand and provide written informed consent prior to participation in this study.
* A female is eligible to enter and participate in the study if she is of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
  2. Child-bearing potential, has a negative pregnancy test at screen and agrees to one of the following methods of contraception (any contraception method must be used consistently and correctly, i.e., in accordance with both the approved product label and the instructions of a physician):

Complete abstinence from intercourse from 2 weeks prior to administration of the investigational products, throughout the study, and for at least 2 weeks after discontinuation of all study medications Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide). Hormonal contraception will not be considered adequate for inclusion into this study Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year.

Sterilization (female subject or male partner of female subject).

* Prior to randomization, subjects must have been screened and be negative for the HLA-B*5701 allele. Test may be performed by local laboratory and results must be available for source document verification according to local practices.

Exclusion Criteria:

* Subject is in the initial acute phase of a CDC Clinical Category C infection at Baseline.
* Subject is enrolled in one or more investigational drug protocols, which may impact HIV RNA suppression.
* Subject is, in the opinion of the Investigator, unable to complete the study dosing period and protocol evaluations and assessments.
* Subject is either pregnant or breastfeeding.
* Subject suffers from a serious medical condition, which in the opinion of the Investigator would compromise the safety of the subject.
* Subject has a history of inflammatory bowel disease or other gastrointestinal dysfunction.
* Subject has any acute laboratory abnormality at screening.
* Subject has an estimated creatinine clearance within the screening period <50mL/min via the Cockcroft-Gault method.
* Alanine aminotransferase (ALT) >5 times the upper limit of normal.
* Subjects with a history of thyroid disease, hyperparathyroid disease, chronic hyper or hypocalcemia, vitamin D deficiency, or receiving thyroid hormone or parathyroid hormone replacement within 28 days prior to screening.
* Subjects with a history of systemic inflammatory arthritis.
* Subjects who are hepatitis B positive at screening.
* Subject requires treatment with radiation therapy or cytotoxic chemotherapeutic agents.
* Subject has received treatment with an HIV-1 immunotherapeutic vaccine or any agents with documented activity against HIV-1 in vitro within 28 days prior to Screening, or an anticipated need during the study.
* Subjects who require treatment with any of the following medications within 28 days of commencement of investigational product, or an anticipated need during the study:
* Medications with significant drug-drug interactions with efavirenz:voriconazole, terfenadine, astemizole, cisapride, ergot alkaloids (dihydroergotamine, ergonovine, ergotamine, methylergonovine), midazolam, triazolam, St. John's wort, carbamazepine, phenytoin, phenobarbital, rifampin, pimozide, bepridil
* Medications which may impact on bone mineral density: oral or systemic corticosteroids, anticonvulsants, heparin, warfarin, cyclosporine, bisphosphonates, calcitonin, parathyroid hormone, Vitamin D supplements and analogues, Calcium supplements, oestrogen or progesterone replacement (oral hormonal contraception permitted), raloxifene, tamoxifen, testosterone or anabolic steroid replacement/supplements.
* Systemic interleukins or interferons
* Subject has a history of allergy to any of the protocol-specified medications or any excipients therein.
* Subject has evidence of genotypic resistance at screening (according to central lab interpretation) or prior documented evidence of genotypic and/or phenotypic (above threshold for reduced susceptibility) resistance to any of the following drugs: efavirenz, abacavir, lamivudine, tenofovir, emtricitabine.
* Subjects who are unsuitable for DEXA scanning should be excluded, including 1) Less than three vertebra in the range of L1 to L4 that are suitable for BMD measurement by DEXA, or 2) Bilateral hip replacement.
* The subject has previously participated in an experimental drug and/or vaccine trial(s) within 60 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine - whichever is longer, prior to screening for the study.
* The subject will participate simultaneously in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (57):
- Austria (3):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Belgium (5):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Denmark (5):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus N
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense C
- France (3):
  - GSK Investigational Site, Garches
  - GSK Investigational Site, Levallois-Perret
  - GSK Investigational Site, Saint-Denis
- Germany (8):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Dublin, Ireland
- Italy (7):
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Legnano (MI, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- GSK Investigational Site, Riga, Latvia
- Netherlands (5):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Utrecht
- GSK Investigational Site, Amadora, Portugal
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- Switzerland (5):
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Sankt Gallen
  - GSK Investigational Site, Zurich
- United Kingdom (11):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Woolwich, London, London
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Brighton, Sussex East
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Farnworth, Bolton
  - GSK Investigational Site, Gloucester
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Background] Post FA, Moyle GJ, Stellbrink HJ, Domingo P, Podzamczer D, Fisher M, Norden AG, Cavassini M, Rieger A, Khuong-Josses MA, Branco T, Pearce HC, Givens N, Vavro C, Lim ML. Randomized comparison of renal effects, efficacy, and safety with once-daily abacavir/lamivudine versus tenofovir/emtricitabine, administered with efavirenz, in antiretroviral-naive, HIV-1-infected adults: 48-week results from the ASSERT study. J Acquir Immune Defic Syndr. 2010 Sep;55(1):49-57. doi: 10.1097/QAI.0b013e3181dd911e. PMID 20431394

RESULTS

PARTICIPANT FLOW:
Groups:
- ABC/3TC FDC: Abacavir (ABC) 600 mg/lamivudine (3TC) 300 mg fixed dose combination (FDC) once daily (QD) plus 600 mg efavirenz QD
- TDF/FTC FDC: Tenofovir (TDF) 300 mg/emtricitabine (FTC) 200 mg FDC once daily (QD) plus 600 mg efavirenz QD
Period: Overall Study
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Started | 195 (Three participants were randomized but were not exposed to study drug (ABC/3TC).) | 197 (Four participants were randomized but were not exposed to study drug (TDF/FTC).)
Completed | 115 | 134
Not Completed | 80 | 63
Not completed — Adverse Event | 28 | 26
Not completed — Insufficient Viral Load Response | 4 | 2
Not completed — Protocol-defined Virological Failure | 7 | 0
Not completed — Non-compliance | 2 | 4
Not completed — Lost to Follow-up | 7 | 8
Not completed — Treatment Eligibility Criteria Not Met | 3 | 0
Not completed — Protocol Violation | 7 | 2
Not completed — Investigator Decision | 4 | 3
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Disease Progression | 1 | 0
Not completed — Participant Moved | 2 | 0
Not completed — Participant not able to perform Week 96 | 1 | 0
Not completed — Participant moved.Week 96 visit, no scan | 1 | 0
Not completed — Prohibited Medication | 1 | 2
Not completed — Participant planning pregnancy | 1 | 0
Not completed — Participant overweight, no scan possible | 1 | 0
Not completed — No scan facilities | 0 | 2
Not completed — Pregnancy | 0 | 3
Not completed — Not Exposed to Study Drug | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABC/3TC FDC | TDF/FTC FDC | Total
Number analyzed (Participants) | 192 | 193 | 385
Age Continuous [Median (Full Range); unit: Years] — The Intent-to-Treat (ITT)-Exposed (E) Population, comprised of all randomized participants who received at least one dose of study medication, was used for all baseline characteristics.
  Years | 38.0 [19 to 70] | 36.0 [18 to 66] | 37.0 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — The Intent-to-Treat (ITT)-Exposed (E) Population, comprised of all randomized participants who received at least one dose of study medication, was used for all baseline characteristics.
  Participants
    Female | 33 | 40 | 73
    Male | 159 | 153 | 312
Race/Ethnicity, Customized [Number; unit: participants] — The Intent-to-Treat (ITT)-Exposed (E) Population, comprised of all randomized participants who received at least one dose of study medication, was used for all baseline characteristics.
  participants
    African American/African Heritage | 26 | 30 | 56
    American Indian or Alaska Native | 11 | 7 | 18
    Asian | 2 | 5 | 7
    White | 153 | 151 | 304

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Estimated Glomerular Filtration Rate (GFR), Calculated by Modification of Diet in Renal Disease (MDRD) Equation, at Week 48
Description: Change from baseline was calculated as the Week 48 value minus the baseline value. GFR is a measure of the rate at which blood is filtered by the kidney. MDRD is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine, age, race, and gender. GFR (mL/min/1.73 m^2) = 175 * (Scr)^-1.154 * (Age)^-0.203 * (0.742 if female) * (1.212 if African American) (conventional units). mL, milliliters; min, minute; m^2, meters squared; Scr, serum creatinine; BMI, body mass index.
Time Frame: Baseline, Week 48
Population: Intent-to-Treat-Exposed (ITT-E) Population: all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Error); unit: milliliters per minute (mL/min)/1.73 m^2
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
milliliters per minute (mL/min)/1.73 m^2 | 0.22 (0.890) | 1.18 (0.828)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.435, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline GFR by MDRD, baseline BMI, race group, treatment*visit, baseline GFR by MDRD*visit and baseline BMI*visit; The correlation matrix for within-subject errors is unstructured

2. Secondary Outcome: Mean Change From Baseline in Estimated Glomerular Filtration Rate (GFR), Calculated by Modification of Diet in Renal Disease (MDRD) Equation, at Week 24
Description: Change from baseline was calculated as the Week 24 value minus the baseline value. GFR is a measure of the rate at which blood is filtered by the kidney. MDRD is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine, age, race, and gender. GFR (mL/min/1.73 m^2) = 175 * (Scr)^-1.154 * (Age)^-0.203 * (0.742 if female) * (1.212 if African American) (conventional units). mL, milliliters; min, minute; m^2, meters squared; Scr, serum creatinine.
Time Frame: Baseline, Week 24
Population: ITT-E Population
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
mL/min/1.73m^2 | 2.78 (0.884) | 0.43 (0.842)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.057, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline GFR by MDRD, baseline BMI, race group, age group, treatment*visit, baseline GFR by MDRD*visit and baseline BMI*visit; The correlation matrix for within-subject errors is unstructured

3. Secondary Outcome: Mean Change From Baseline in Estimated Glomerular Filtration Rate (GFR), Calculated by Modification of Diet in Renal Disease (MDRD) Equation, at Week 96
Description: Change from baseline was calculated as the Week 96 value minus the baseline value. GFR is a measure of the rate at which blood is filtered by the kidney. MDRD is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine, age, race, and gender. GFR (mL/min/1.73 m^2) = 175 * (Scr)^-1.154 * (Age)^-0.203 * (0.742 if female) * (1.212 if African American) (conventional units). mL, milliliters; min, minute; m^s, meters squared; Scr, serum creatinine.
Time Frame: Baseline, Week 96
Population: ITT-E Population
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
mL/min/1.73m^2 | 1.48 (1.022) | -1.15 (0.944)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.060, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The correlation matrix for within-subject errors is unstructured

4. Secondary Outcome: Mean Change From Baseline in Estimated GFR, Calculated by Cockcroft-Gault Equation, at Week 24
Description: Change from baseline was calculated as the Week 24 value minus the baseline value. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. GFR = (140 - age) * (mass in kg) * (0.85 if female) divided by 72 * serum creatinine in mg/dL. mg, milligram; dL, deciliter; kg, kilogram; CG, Cockcroft-Gault.
Time Frame: Baseline, Week 24
Population: ITT-E Population
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
mL/min | 4.27 (0.944) | 2.54 (0.897)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.186, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline GFR by CG, baseline BMI, race group, age group, hypertension, treatment*visit, baseline GFR by CG*visit and baseline BMI*visit; The correlation matrix for within-subject errors is unstructured

5. Secondary Outcome: Mean Change From Baseline in Estimated GFR, Calculated by Cockcroft-Gault Equation, at Week 48
Description: Change from baseline was calculated as the Week 48 value minus the baseline value. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. GFR = (140 - age) * (mass in kg) * (0.85 if female) divided by 72 * serum creatinine in mg/dL. mg, milligram; dL, deciliter; kg, kilogram.
Time Frame: Baseline, Week 48
Population: ITT-E Population
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
mL/min | 2.66 (1.005) | 3.80 (0.933)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.413, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; The correlation matrix for within-subject errors is unstructured

6. Secondary Outcome: Mean Change From Baseline in Estimated GFR, Calculated by Cockcroft-Gault Equation, at Week 96
Description: Change from baseline was calculated as the Week 96 value minus the baseline value. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. GFR = (140 - age) * (mass in kg) * (0.85 if female) divided by 72 * serum creatinine in mg/dL. mg, milligram; dL, deciliter; kg, kilogram.
Time Frame: Baseline, Week 96
Population: ITT-E Population
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
mL/min | 4.37 (1.228) | 2.68 (1.133)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.315, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline GFR by CG, baseline BMI, race group, baseline CD4, treatment*visit, baseline GFR by CG*visit, baseline BMI*visit and baseline CD4*visit; The correlation matrix for within-subject errors is unstructured

7. Secondary Outcome: Number of Participants With Decline From Baseline in Estimated GFR, Calculated by MDRD and Cockcroft-Gault Equations, of >=10 mL/Min/1.73 m^2 (mL/Min for Cockcroft-Gault), >=20 mL/Min/1.72 m^2, >=10%, and >=20% at Week 24
Description: mL, milliliter; min, minute; m^2, meters squared
Time Frame: Baseline, Week 24
Population: ITT-E Population. Some participants had withdrawn from the study by Week 24.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 156 | 173
participants
  >=10 mL/min, MDRD | 16 | 26
  >=10 mL/min, Cockcroft-Gault | 16 | 20
  >=20 mL/min, MDRD | 4 | 6
  >=20 mL/min, Cockcroft-Gault | 3 | 4
  >=10%, MDRD | 15 | 24
  >=10%, Cockcroft-Gault | 10 | 17
  >=20%, MDRD | 2 | 3
  >=20%, Cockcroft-Gault | 2 | 3

8. Secondary Outcome: Number of Participants With Decline From Baseline in Estimated GFR, Calculated by MDRD and Cockcroft-Gault Equations, of >=10 mL/Min/1.73m^2 (mL/Min for Cockcroft-Gault), >=20 mL/Min/1.72m^2, >=10%, and >=20% at Week 48
Description: mL, milliliter; min, minute; m^2, meters squared
Time Frame: Baseline, Week 48
Population: ITT-E Population. Some participants had withdrawn by Week 48.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 136 | 159
participants
  >=10 mL/min, MDRD | 23 | 21
  >=10 mL/min, Cockcroft-Gault | 15 | 14
  >=20 mL/min, MDRD | 4 | 3
  >=20 mL/min, Cockcroft-Gault | 4 | 2
  >=10%, MDRD | 21 | 21
  >=10%, Cockcroft-Gault | 11 | 9
  >=20%, MDRD | 4 | 2
  >=20%, Cockcroft-Gault | 3 | 0

9. Secondary Outcome: Number of Participants With Decline From Baseline in Estimated GFR, Calculated by MDRD and Cockcroft-Gault Equations, of >=10 mL/Min/1.73m^2 (mL/Min for Cockcroft-Gault), >=20 mL/Min/1.72m^2, >=10%, and >=20% at Week 96
Description: mL, milliliter; min, minute; m^2, meters squared
Time Frame: Baseline, Week 96
Population: ITT-E Population. Some participants had withdrawn by Week 96.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 111 | 131
participants
  >=10 mL/min, MDRD | 15 | 38
  >=10 mL/min, Cockcroft-Gault | 11 | 19
  >=20 mL/min, MDRD | 4 | 7
  >=20 mL/min, Cockcroft-Gault | 4 | 5
  >=10%, MDRD | 15 | 27
  >=10%, Cockcroft-Gault | 12 | 16
  >=20%, MDRD | 3 | 6
  >=20%, Cockcroft-Gault | 3 | 4

10. Secondary Outcome: Number of Participants With National Kidney Foundation Chronic Kidney Disease Stage 1, 2, 3, 4, or 5 Categories of Renal Function at Week 24
Description: Normal: GFR >=60 mL/min/1.73 m^2 and creatinine ratio <=200 mg/g GFR; Stage 1: GFR >=90 mL/min/1.73 m^2 and creatinine ratio >200 mg/g; Stage 2: GFR >=60-<90 mL/min/1.73 m^2 and creatinine ratio >200 mg/g; Stage 3: GFR >=30-<60 mL/min/1.73 m^2; Stage 4: GFR >=15-<30 mL/min/1.73 m^2; Stage 5: GFR <15 mL/min/1.73 m^2. mL, milliliter; min, minute; m^2, meters squared; mg, milligram; g, gram.
Time Frame: Baseline, Week 24
Population: ITT-E Population. Some participants had withdrawn by Week 24.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 114 | 135
participants
  Normal | 97 | 114
  Stage 1 | 11 | 15
  Stage 2 | 5 | 5
  Stage 3 | 1 | 1
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

11. Secondary Outcome: Number of Participants With National Kidney Foundation Chronic Kidney Disease Stage 1, 2, 3, 4, or 5 Categories of Renal Function at Week 48
Description: as for outcome 10
Time Frame: Baseline, Week 48
Population: ITT-E Population. Some participants had withdrawn by Week 48.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 112 | 133
participants
  Missing | 12 | 19
  Normal | 90 | 106
  Stage 1 | 7 | 5
  Stage 2 | 3 | 3
  Stage 3 | 0 | 0
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

12. Secondary Outcome: Number of Participants With National Kidney Foundation Chronic Kidney Disease Stage 1, 2, 3, 4, or 5 Categories of Renal Function at Week 96
Description: as for outcome 10
Time Frame: Baseline, Week 96
Population: ITT-E Population. Some participants had withdrawn by Week 96.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 93 | 109
participants
  Missing | 11 | 18
  Normal | 75 | 83
  Stage 1 | 3 | 4
  Stage 2 | 4 | 4
  Stage 3 | 0 | 0
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

13. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD), Measured by Dual-energy X-ray Absorptiometry (DXA), at Week 24
Description: BMD is a measure (grams [g] per centimeters cubed [cm^3]) of the mineral content of bone in a particular skeletal area. DXA scans use low energy x-rays to measure the density of bones. The standard error (SE) of both treatment groups was based on the model on the log scale.
Time Frame: Baseline, Week 24
Population: ITT-E Population
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
percent change | -2.12 (0.0011) | -3.30 (0.0011)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline spine BMD, baseline BMI, race group, age group, hypertension, treatment*visit, baseline spine BMD*visit and baseline BMI*visit; The correlation matrix for within-subject errors is unstructured

14. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD), Measured by Dual-energy X-ray Absorptiometry (DXA), at Week 24
Description: BMD is a measure (grams per cm^3) of the mineral content of bone in a particular skeletal area. DXA scans use low energy x-rays to measure the density of bones. The standard error (SE) of both treatment groups was based on the model on the log scale.
Time Frame: Baseline, Week 24
Population: ITT-E Population
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
percent change | -1.19 (0.0007) | -2.73 (0.0007)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline hip BMD, baseline BMI, race group, risk factor, country group, treatment*visit, baseline hip BMD*visit and baseline BMI*visit; The correlation matrix for within-subject errors is unstructured

15. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD), Measured by Dual-energy X-ray Absorptiometry (DXA), at Week 48
Description: as for outcome 14
Time Frame: Baseline, Week 48
Population: ITT-E Population
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
percent change | -1.59 (0.0013) | -2.41 (0.0012)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline spine BMD, baseline BMI, race group, age group, treatment*visit, baseline spine BMD*visit and baseline BMI*visit; The correlation matrix for within-subject errors is unstructured

16. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD), Measured by Dual-energy X-ray Absorptiometry (DXA), at Week 48
Description: as for outcome 14
Time Frame: Baseline, Week 48
Population: ITT-E Population
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
percent change | -1.90 (0.0010) | -3.56 (0.0009)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline hip BMD, baseline BMI, race group, risk factor, prohibited medication, previous fracture, treatment*visit, baseline hip BMD*visit and baseline BMI*visit; Correlation matrix for within-subject errors is unstructured

17. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD), Measured by Dual-energy X-ray Absorptiometry (DXA), at Week 96
Description: as for outcome 14
Time Frame: Baseline, Week 96
Population: ITT-E Population
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
percent change | -0.87 (0.0017) | -1.70 (0.0015)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.112, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]; correlation matrix for within-subject errors is unstructured

18. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD), Measured by Dual-energy X-ray Absorptiometry (DXA), at Week 96
Description: as for outcome 14
Time Frame: Baseline, Week 96
Population: ITT-E Population
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
percent change | -2.17 (0.0013) | -3.55 (0.0012)
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The model includes the following covariates: treatment, visit, baseline hip BMD, baseline BMI, race group, risk factor, prohibited medication, previous fracture, treatment*visit, baseline hip BMD*visit, and baseline BMI*visit; The correlation matrix for within-subject errors is unstructured

19. Secondary Outcome: Number of Participants With a Decline From Baseline in Lumbar Spine and Hip Bone Mineral Density (BMD) >=2.0% and >=6.0% at Week 24
Description: BMD is a measure of the mineral content of bone in a particular skeletal area. DXA scans use low energy x-rays to measure the density of bones.
Time Frame: Baseline, Week 24
Population: ITT-E Population. Some participants had withdrawn by Week 24/did not have a DXA scan performed. DXA, dual energy x-ray absorptiometry.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 142 | 165
participants
  >=2%, spine, n=142, 165 | 73 | 115
  >=6%, spine, n=142, 165 | 10 | 17
  >=2%, hip, n=137, 160 | 38 | 93
  >=6%, hip, n=137, 160 | 1 | 6

20. Secondary Outcome: Number of Participants With a Decline From Baseline in Lumbar Spine and Hip Bone Mineral Density (BMD) >=2.0% and >=6.0% at Week 48
Description: as for outcome 19
Time Frame: Baseline, Week 48
Population: ITT-E Population. Some participants had withdrawn by Week 48/did not have a DXA scan performed. DXA, dual energy x-ray absorptiometry.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 125 | 141
participants
  >=2%, spine, n=125, 141 | 51 | 84
  >=6%, spine, n=125, 141 | 5 | 13
  >=2%, hip, n=119, 140 | 54 | 111
  >=6%, hip, n=119, 140 | 3 | 17

21. Secondary Outcome: Number of Participants With a Decline From Baseline in Lumbar Spine and Hip Bone Mineral Density (BMD) >=2.0% and >=6.0% at Week 96
Description: as for outcome 19
Time Frame: Baseline, Week 96
Population: ITT-E Population. Some participants had withdrawn by Week 96/did not have a DXA scan performed. DXA, dual energy x-ray absorptiometry.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 59 | 79
participants
  >=2%, spine, n=59, 79 | 21 | 39
  >=6%, spine, n=59, 79 | 3 | 8
  >=2%, hip, n=58, 76 | 33 | 52
  >=6%, hip, n=58, 76 | 1 | 13

22. Secondary Outcome: Number of Participants Meeting World Health Organization (WHO) Criteria for Osteopenia (T-score of -2.5 to -1.0) and Osteoporosis (T-score of <-2.5) at Week 24
Description: The T-score is a radiographic diagnosis that compares bone mineral density (BMD) to that of a "normal, healthy, 30-year-old female". The lower the T-score, the lower the BMD. A T-score of +1 to -1 is normal. A T-score decrease of -1 indicates a 10%-15% decrease in BMD.
Time Frame: Week 24
Population: ITT-E Population. Some participants had withdrawn by Week 24.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 149 | 173
participants
  Osteopenia, spine, n=147, 173 | 41 | 68
  Osteporosis, spine, n=147, 173 | 16 | 9
  Osteopenia, hip, n=149, 170 | 38 | 54
  Osteoporosis, hip, n=149, 170 | 4 | 1

23. Secondary Outcome: Number of Participants Meeting World Health Organization (WHO) Criteria for Osteopenia (T-score of -2.5 to -1.0) and Osteoporosis (T-score of <-2.5) at Week 48
Description: as for outcome 22
Time Frame: Week 48
Population: ITT-E Population. Some participants had withdrawn by Week 48.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 132 | 147
participants
  Osteopenia, spine, n=132, 147 | 41 | 57
  Osteporosis, spine, n=132, 147 | 15 | 5
  Osteopenia, hip, n=130, 147 | 37 | 50
  Osteoporosis, hip, n=130, 147 | 4 | 0

24. Secondary Outcome: Number of Participants Meeting World Health Organization (WHO) Criteria for Osteopenia (T-score of -2.5 to -1.0) and Osteoporosis (T-score of <-2.5) at Week 96
Description: as for outcome 22
Time Frame: Week 96
Population: ITT-E Population. Some participants had withdrawn by Week 96.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 65 | 82
participants
  Osteopenia, spine, n=64, 82 | 21 | 34
  Osteporosis, spine, n=64, 82 | 5 | 3
  Osteopenia, hip, n=65, 80 | 20 | 31
  Osteoporosis, hip, n=65, 80 | 0 | 0

25. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE) Leading to Discontinuation by Week 24
Description: An adverse event was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events occurring in two or more participants are presented.
Time Frame: Baseline to Week 24
Population: Safety Population: all randomized participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Any event | 26 | 14
  Drug hypersensitivity | 11 | 1
  Rash | 2 | 3
  Dizziness | 0 | 2
  Hypersensitivity | 3 | 0
  Drug eruption | 1 | 1

26. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE) Leading to Discontinuation by Week 48
Description: as for outcome 25
Time Frame: Baseline to Week 48
Population: Safety Population: all randomized participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Any event | 29 | 21
  Drug hypersensitivity | 11 | 1
  Bone density decreased | 0 | 2
  Rash | 2 | 3
  Dizziness | 1 | 3
  Hypersensitivity | 3 | 0
  Drug eruption | 1 | 1

27. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE) Leading to Discontinuation by Week 96
Description: as for outcome 25
Time Frame: Baseline to Week 96
Population: Safety Population: all randomized participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Any event | 33 | 28
  Drug hypersensitivity | 11 | 1
  Bone density decreased | 0 | 8
  Rash | 2 | 3
  Dizziness | 1 | 3
  Hypersensitivity | 3 | 0
  Abnormal dreams | 3 | 0
  Drug eruption | 1 | 1
  Depression | 0 | 2

28. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting Total Cholesterol at Week 24
Description: Blood samples were collected from participants for analysis of their lipid profile. Data are categorized by the maximum post-baseline threshold reached. <200 mg/dL, desirable; 200-<240 mg/dL, borderline high; >=240 mg/dL, high. mg, milligram; dL, deciliter.
Time Frame: Baseline, Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Desirable to desirable | 54 | 104
  Desirable to borderline high | 47 | 29
  Desirable to high | 32 | 9
  Borderline high to desirable | 1 | 3
  Borderline high to borderline high | 2 | 9
  Borderline high to high | 10 | 6
  High to desirable | 0 | 0
  High to borderline high | 0 | 0
  High to high | 3 | 2

29. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting Total Cholesterol at Week 48
Description: as for outcome 28
Time Frame: Baseline, Week 48
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Desirable to desirable | 46 | 96
  Desirable to borderline high | 52 | 37
  Desirable to high | 36 | 9
  Borderline high to desirable | 1 | 1
  Borderline high to borderline high | 2 | 9
  Borderline high to high | 10 | 8
  High to desirable | 0 | 0
  High to borderline high | 0 | 0
  High to high | 3 | 2

30. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting Total Cholesterol at Week 96
Description: as for outcome 28
Time Frame: Baseline, Week 96
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Desirable to desirable | 39 | 86
  Desirable to borderline high | 49 | 47
  Desirable to high | 46 | 10
  Borderline high to desirable | 1 | 1
  Borderline high to borderline high | 2 | 9
  Borderline high to high | 10 | 8
  High to desirable | 0 | 0
  High to borderline high | 0 | 0
  High to high | 3 | 2

31. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Low-density Lipoprotein (LDL) at Week 24
Description: Blood samples were collected from participants for analysis of their lipid profile. Data are categorized by the maximum post-baseline threshold reached. <100 mg/dL, optimal; 100-<130 mg/dL, near/above optimal; 130-<160 mg/dL, borderline high; 160-<190 mg/dL, high; >=190 mg/dL, very high.
Time Frame: Baseline, Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Optimal to optimal | 22 | 46
  Optimal to near or above optimal | 41 | 43
  Optimal to borderline high | 22 | 11
  Optimal to high | 6 | 1
  Optimal to very high | 1 | 0
  Near or above optimal to optimal | 0 | 5
  Near or above optimal to near or above optimal | 6 | 22
  Near or above optimal to borderline high | 17 | 11
  Near or above optimal to high | 12 | 5
  Near or above optimal to very high | 4 | 1
  Borderline high to optimal | 0 | 0
  Borderline high to near or above optimal | 1 | 6
  Borderline high to borderline high | 2 | 3
  Borderline high to high | 4 | 3
  Borderline high to very high | 3 | 2
  High to optimal | 0 | 0
  High to near or above optimal | 0 | 0
  High to borderline high | 0 | 0
  High to high | 1 | 1
  High to very high | 0 | 0
  Very high to optimal | 0 | 0
  Very high to near or above optimal | 0 | 0
  Very high to borderline high | 1 | 0
  Very high to high | 0 | 0
  Very high to very high | 1 | 1

32. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Low-density Lipoprotein (LDL) at Week 48
Description: as for outcome 31
Time Frame: Baseline, Week 48
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Optimal to optimal | 20 | 42
  Optimal to near or above optimal | 38 | 46
  Optimal to borderline high | 27 | 12
  Optimal to high | 8 | 1
  Optimal to very high | 1 | 0
  Near or above optimal to optimal | 0 | 3
  Near or above optimal to near or above optimal | 4 | 21
  Near or above optimal to borderline high | 19 | 13
  Near or above optimal to high | 12 | 6
  Near or above optimal to very high | 4 | 1
  Borderline high to optimal | 0 | 0
  Borderline high to near or above optimal | 1 | 3
  Borderline high to borderline high | 2 | 5
  Borderline high to high | 3 | 4
  Borderline high to very high | 4 | 2
  High to optimal | 0 | 0
  High to near or above optimal | 0 | 0
  High to borderline high | 0 | 0
  High to high | 1 | 1
  High to very high | 0 | 0
  Very high to optimal | 0 | 0
  Very high to near or above optimal | 0 | 0
  Very high to borderline high | 1 | 0
  Very high to high | 0 | 0
  Very high to very high | 1 | 1

33. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Low-density Lipoprotein (LDL) at Week 96
Description: as for outcome 31
Time Frame: Baseline, Week 96
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Optimal to optimal | 18 | 37
  Optimal to near or above optimal | 35 | 46
  Optimal to borderline high | 29 | 17
  Optimal to high | 9 | 1
  Optimal to very high | 3 | 0
  Near or above optimal to optimal | 0 | 1
  Near or above optimal to near or above optimal | 4 | 19
  Near or above optimal to borderline high | 17 | 16
  Near or above optimal to high | 12 | 7
  Near or above optimal to very high | 6 | 2
  Borderline high to optimal | 0 | 0
  Borderline high to near or above optimal | 1 | 3
  Borderline high to borderline high | 2 | 5
  Borderline high to high | 3 | 3
  Borderline high to very high | 4 | 3
  High to optimal | 0 | 0
  High to near or above optimal | 0 | 0
  High to borderline high | 0 | 0
  High to high | 1 | 1
  High to very high | 0 | 0
  Very high to optimal | 0 | 0
  Very high to near or above optimal | 0 | 0
  Very high to borderline high | 1 | 0
  Very high to high | 0 | 0
  Very high to very high | 1 | 1

34. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting High-density Lipoprotein (HDL) at Week 24
Description: Blood samples were collected from participants for analysis of their lipid profile. Data are categorized by the maximum post-baseline threshold reached. <40 mg/dL, low; 40-<60 mg/dL, normal; >=60 mg/dL, high.
Time Frame: Baseline, Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Low to low | 19 | 36
  Low to normal | 72 | 66
  Low to high | 10 | 9
  Normal to low | 0 | 1
  Normal to normal | 12 | 30
  Normal to high | 26 | 12
  High to low | 0 | 0
  High to normal | 0 | 3
  High to high | 10 | 5

35. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting High-density Lipoprotein (HDL) at Week 48
Description: as for outcome 34
Time Frame: Baseline, Week 48
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Low to low | 17 | 28
  Low to normal | 67 | 73
  Low to high | 18 | 10
  Normal to low | 0 | 0
  Normal to normal | 11 | 23
  Normal to high | 27 | 20
  High to low | 0 | 0
  High to normal | 0 | 3
  High to high | 10 | 5

36. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting High-density Lipoprotein (HDL) at Week 96
Description: as for outcome 34
Time Frame: Baseline, Week 96
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Low to low | 11 | 23
  Low to normal | 66 | 75
  Low to high | 25 | 13
  Normal to low | 0 | 0
  Normal to normal | 8 | 17
  Normal to high | 30 | 27
  High to low | 0 | 0
  High to normal | 0 | 1
  High to high | 10 | 7

37. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting Triglycerides at Week 24
Description: Blood samples were collected from participants for analysis of their lipid profile. Data are categorized by the maximum post-baseline threshold reached. <150 mg/dL, normal; 150-<200 mg/dL, borderline high; 200-<500 mg/dL, high; >=500 mg/dL, very high.
Time Frame: Baseline, Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Normal to normal | 63 | 78
  Normal to borderline high | 21 | 19
  Normal to high | 23 | 9
  Normal to very high | 0 | 0
  Borderline high to normal | 5 | 7
  Borderline high to borderline high | 5 | 10
  Borderline high to high | 9 | 15
  Borderline high to very high | 0 | 0
  High to normal | 2 | 6
  High to borderline high | 5 | 3
  High to high | 12 | 15
  High to very high | 3 | 0
  Very high to normal | 0 | 0
  Very high to borderline high | 0 | 0
  Very high to high | 0 | 1
  Very high to very high | 1 | 0

38. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting Triglycerides at Week 48
Description: as for outcome 37
Time Frame: Baseline, Week 48
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Normal to normal | 55 | 70
  Normal to borderline high | 22 | 23
  Normal to high | 30 | 12
  Normal to very high | 0 | 1
  Borderline high to normal | 4 | 6
  Borderline high to borderline high | 5 | 7
  Borderline high to high | 11 | 19
  Borderline high to very high | 0 | 0
  High to normal | 2 | 5
  High to borderline high | 4 | 3
  High to high | 12 | 15
  High to very high | 4 | 0
  Very high to normal | 0 | 0
  Very high to borderline high | 0 | 0
  Very high to high | 0 | 1
  Very high to very high | 1 | 0

39. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in National Cholesterol Education Program (NCEP) Thresholds for Fasting Triglycerides at Week 96
Description: Blood samples were collected from participants for analysis of their lipid profile. Data are categorized by the maximum post-baseline threshold reached. <150 mg/dL, normal; 150->200 mg/dL, borderline high; 200-<500 mg/dL, high;>= 500 mg/dL, very high.
Time Frame: Baseline, Week 96
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Normal to normal | 47 | 55
  Normal to borderline high | 25 | 31
  Normal to high | 34 | 20
  Normal to very high | 1 | 1
  Borderline high to normal | 4 | 5
  Borderline high to borderline high | 4 | 8
  Borderline high to high | 11 | 19
  Borderline high to very high | 1 | 0
  High to normal | 2 | 5
  High to borderline high | 4 | 2
  High to high | 11 | 16
  High to very high | 5 | 0
  Very high to normal | 0 | 0
  Very high to borderline high | 0 | 0
  Very high to high | 0 | 1
  Very high to very high | 1 | 0

40. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Division of AIDS (DAIDS) Toxicities at Week 24
Description: The DAIDS toxicity table provides descriptive terminology for grading the severity of adult adverse events. Laboratory grades also provide ranges for each parameter. Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: potentially life-threatening. LDL, low-density lipid; HDL, high-density lipid. Treatment emergent refers to any toxicity that was not present prior to the start of study drug treatment.
Time Frame: Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Cholesterol, Grade 3 | 6 | 1
  Cholesterol, Grade 4 | 0 | 0
  LDL cholesterol, Grade 3 | 8 | 3
  LDL cholesterol, Grade 4 | 0 | 0
  Non-HDL cholesterol, Grade 3 | 19 | 5
  Non-HDL cholesterol, Grade 4 | 0 | 0
  Triglycerides, Grade 3 | 2 | 0
  Triglycerides, Grade 4 | 0 | 0
  Alanine aminotransferase, Grade 3 | 1 | 3
  Alanine aminotransferase, Grade 4 | 1 | 1
  Aspartate aminotransferase, Grade 3 | 1 | 0
  Aspartate aminotransferase, Grade 4 | 1 | 2
  Alkaline phosphatase, Grade 3 | 0 | 1
  Alkaline phosphatase, Grade 4 | 0 | 0
  Creatinine kinase, Grade 3 | 0 | 1
  Creatinine kinase, Grade 4 | 1 | 1
  Phosphorus inorganic, Grade 3 | 1 | 1
  Phosphorus inorganic, Grade 4 | 0 | 0
  Lipase, Grade 3 | 3 | 1
  Lipase, Grade 4 | 2 | 0
  Hyperkalaemia, Grade 3 | 0 | 0
  Hyperkalaemia, Grade 4 | 1 | 1
  Glomerular filtration rate, MDRD, Grade 3 | 1 | 1
  Glomerular filtration rate, MDRD, Grade 4 | 0 | 0
  Total neutrophils, Grade 3 | 1 | 0
  Total neutrophils, Grade 4 | 1 | 2
  Thrombocytopenia, Grade 3 | 1 | 0
  Thrombocytopenia, Grade 4 | 0 | 0

41. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Division of AIDS (DAIDS) Toxicities at Week 48
Description: as for outcome 40
Time Frame: Week 48
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Cholesterol, Grade 3 | 7 | 1
  Cholesterol, Grade 4 | 0 | 0
  LDL cholesterol, Grade 3 | 9 | 3
  LDL cholesterol, Grade 4 | 0 | 0
  Non-HDL cholesterol, Grade 3 | 20 | 6
  Non-HDL cholesterol, Grade 4 | 0 | 0
  Triglycerides, Grade 3 | 3 | 0
  Triglycerides, Grade 4 | 0 | 0
  Alanine aminotransferase, Grade 3 | 2 | 4
  Alanine aminotransferase, Grade 4 | 2 | 1
  Aspartate aminotransferase, Grade 3 | 2 | 0
  Aspartate aminotransferase, Grade 4 | 2 | 2
  Alkaline phosphatase, Grade 3 | 0 | 1
  Alkaline phosphatase, Grade 4 | 0 | 0
  Total bilirubin Grade 3 | 1 | 0
  Total bilirubin, Grade 4 | 0 | 0
  Creatinine kinase, Grade 3 | 0 | 2
  Creatinine kinase, Grade 4 | 1 | 1
  Phosphorus inorganic, Grade 3 | 3 | 1
  Phosphorus inorganic, Grade 4 | 0 | 0
  Lipase, Grade 3 | 5 | 1
  Lipase, Grade 4 | 2 | 0
  Hyperkalaemia, Grade 3 | 0 | 0
  Hyperkalaemia, Grade 4 | 2 | 2
  Glomerular filtration rate, MDRD, Grade 3 | 1 | 1
  Glomerular filtration rate, MDRD, Grade 4 | 0 | 0
  Total neutrophils, Grade 3 | 2 | 0
  Total neutrophils, Grade 4 | 3 | 2
  Thrombocytopenia, Grade 4 | 1 | 0
  Thrombocytopenia, Grade 4 | 0 | 0

42. Secondary Outcome: Number of Participants With the Indicated Treatment-emergent Division of AIDS (DAIDS) Toxicities at Week 96
Description: The DAIDS toxicity table provides descriptive terminology for grading the severity of adult adverse events. Laboratory grades also provide ranges for each parameter. Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: potentially life-threatening. LDL, low-density lipid; HDL, high-density lipid. Treatment emergent refers to any toxicity that was not present prior to the start of study drug therapy.
Time Frame: Week 96
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  Cholesterol, Grade 3 | 9 | 1
  Cholesterol, Grade 4 | 0 | 0
  LDL cholesterol, Grade 3 | 13 | 5
  LDL cholesterol, Grade 4 | 0 | 0
  Non-HDL cholesterol, Grade 3 | 22 | 5
  Non-HDL cholesterol, Grade 4 | 0 | 0
  Triglycerides, Grade 3 | 2 | 0
  Triglycerides, Grade 4 | 1 | 0
  Alanine aminotransferase, Grade 3 | 2 | 4
  Alanine aminotransferase, Grade 4 | 2 | 1
  Aspartate aminotransferase, Grade 3 | 2 | 1
  Aspartate aminotransferase, Grade 4 | 2 | 2
  Alkaline phosphatase, Grade 3 | 0 | 1
  Alkaline phosphatase, Grade 4 | 0 | 0
  Total bilirubin, Grade 3 | 1 | 0
  Total bilirubin, Grade 4 | 0 | 0
  Creatinine kinase, Grade 3 | 0 | 2
  Creatinine kinase, Grade 4 | 1 | 2
  Phosphorus inorganic, Grade 3 | 4 | 3
  Phosphorus inorganic, Grade 4 | 0 | 0
  Lipase, Grade 3 | 6 | 2
  Lipase, Grade 4 | 4 | 2
  Hyperkalaemia, Grade 3 | 0 | 0
  Hyperkalaemia, Grade 4 | 2 | 0
  Glomerular filtration rate, MDRD, Grade 3 | 1 | 1
  Glomerular filtration rate, MDRD, Grade 4 | 0 | 0
  Total neutrophils, Grade 3 | 3 | 1
  Total neutrophils, Grade 4 | 5 | 3
  Thrombocytopenia, Grade 3 | 1 | 0
  Thrombocytopenia, Grade 4 | 0 | 0

43. Secondary Outcome: Number of Participants With HIV-1 RNA <50 Copies/Milliliter (c/mL) and 400 c/mL at Week 24
Description: HIV-1 RNA level (viral load) is a strong predictor of the rate of HIV disease progression. It was measured from plasma (participant blood samples) taken at all visits throughout the study. HIV, human immunodeficiency virus; RNA, ribonucleic acid. Viral load is a measure of the severity of the HIV infection.
Time Frame: Week 24
Population: ITT-E Population. Failures and missing values are derived according to the Time to Loss of Virologic Response (TLOVR) Food and Drug Administration (FDA) algorithm.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  <50 copies/mL | 126 | 144
  <400 copies/mL | 147 | 168

44. Secondary Outcome: Number of Participants With HIV-1 RNA <50 Copies/Milliliter (c/mL) and 400 c/mL at Week 48
Description: as for outcome 43
Time Frame: Week 48
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  <50 copies/mL | 121 | 145
  <400 copies/mL | 130 | 151

45. Secondary Outcome: Number of Participants With HIV-1 RNA <50 Copies/Milliliter (c/mL) and 400 c/mL at Week 96
Description: as for outcome 43
Time Frame: Week 96
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 192 | 193
participants
  <50 copies/mL | 98 | 113
  <400 copies/mL | 110 | 126

46. Secondary Outcome: Change From Baseline in Cluster Difference 4 (CD4+) Cell Count at Week 24
Description: CD4+ counts are used to monitor the progression of HIV disease and the strength of the immune system. The number of CD4+ cells decreases as HIV disease progresses. Cell counts were measured from participant blood samples taken throughout the study.
Time Frame: Baseline, Week 24
Population: ITT-E Population. Some participants had withdrawn by Week 24.
Measure: Median (Inter-Quartile Range); unit: cells/millimeters cubed (mm^3)
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 153 | 172
cells/millimeters cubed (mm^3) | 110.0 [50.0 to 180.0] | 100.0 [45.0 to 150.0]

47. Secondary Outcome: Change From Baseline in Cluster Difference 4 (CD4+) Cell Count at Week 48
Description: as for outcome 46
Time Frame: Baseline, Week 48
Population: ITT-E Population. Some participants had withdrawn by Week 48.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 136 | 156
cells/mm^3 | 150.0 [95.0 to 270.0] | 150.0 [80.0 to 215.0]

48. Secondary Outcome: Change From Baseline in Cluster Difference 4 (CD4+) Cell Count at Week 96
Description: as for outcome 46
Time Frame: Baseline, Week 96
Population: ITT-E Population. Some participants had withdrawn by Week 96.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 110 | 128
cells/mm^3 | 235.0 [130.0 to 390.0] | 220.0 [150.0 to 315.0]

49. Secondary Outcome: Number of Participants Classified as Protocol-defined Failures With Treatment-emergent Resistance to Study Drug in the Indicated Viruses at Week 96
Description: Viral resistance was measured using blood samples collected from participants throughout the study. NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor. Virological failure was defined as any one of: participant does not achieve a 1 log10 copies (cop)/mL decrease in plasma HIV-1 RNA by Week (Wk) 4, or has two consecutive plasma HIV-1 RNA measures >=400 cop/mL separated by at least 2-4 wk after being previously <=400 cop/mL on/after Wk 4, or has two consecutive plasma HIV-1 RNA measures >400 cop/mL separated by at least 2-4 wk on/after Wk 24.
Time Frame: Week 96
Population: On-Treatment Resistance: all participants who fulfilled the definition of protocol-defined virological failure (VF) who had paired baseline and VF genotypic data for analysis. One ABC/3TC participant took prohibited medication that potentially lowered efavirenz levels just prior to VF, allowing for the emergence of unexpected NRTI resistance.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 7 | 3
participants
  Any treatment-emergent mutation | 4 | 0
  NRTI | 4 | 0
  NNRTI | 2 | 0

50. Secondary Outcome: Number of Participants Who Indicated "Yes" or "No" to the Question of Whether Unplanned Healthcare Resources Were Utilized
Description: Participants were asked at each visit whether or not they utilized unplanned healthcare resources.
Time Frame: Baseline to Week 96
Population: ITT-E Population. The number of participants analyzed differed by visit because some had withdrawn during the study and some did not have an assessment performed.
Measure: Number; unit: participants
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 178 | 183
participants
  Week 4, Yes, n=178, 183 | 60 | 49
  Week 4, No, n=178, 183 | 118 | 134
  Week 12, Yes, n=162, 177 | 56 | 47
  Week 12, No, n=162, 177 | 106 | 130
  Week 24, Yes, n=156, 173 | 70 | 59
  Week 24, No, n=156, 173 | 86 | 114
  Week 36, Yes, n=148, 169 | 48 | 50
  Week 36, No, n=148, 169 | 100 | 119
  Week 48, Yes, n=137, 161 | 44 | 36
  Week 48, No, n=137, 161 | 93 | 125
  Week 60, Yes, n=129, 148 | 47 | 44
  Week 60, No, n=129, 148 | 82 | 104
  Week 72, Yes, n=126, 139 | 48 | 40
  Week 72, No, n=126, 139 | 78 | 99
  Week 84, Yes, n=121, 136 | 34 | 24
  Week 84, No, n=121, 136 | 87 | 108
  Week 96, Yes, n=113, 135 | 30 | 17
  Week 96, No, n=113, 135 | 83 | 118

51. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in Albumin as a Ratio to Urine Creatinine at Week 96
Description: Renal biomarkers were analyzed using urine samples collected from participants at baseline and Week 96. Renal biomarkers may be an indicator of various aspects of kidney function. The ratio was calculated by dividing the change from baseline albumin value by the urine creatinine value. Albumin is measured in milligrams per millimole (mg/mmol).
Time Frame: Baseline, Week 96
Population: Safety Biomarker Population: all randomized participants who received at least one dose of study medication and had at least one parameter measured at Baseline and at least one post-baseline visit. Some participants had withdrawn by Week 96.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 103 | 120
ratio | 0.872 [0.716 to 1.062] | 0.973 [0.806 to 1.174]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.3025, ANOVA — The model includes the following covariates: treatment, age, baseline biomarker value, and gender; Estimates are calculated from an ANOVA model. Parameters are analyzed based on log transformed data

52. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in Beta 2 Microglobulin (B2M) as a Ratio to Urine Creatinine at Week 96
Description: Renal biomarkers were analyzed using urine samples collected from participants at baseline and Week 96. Renal biomarkers may be an indicator of various aspects of kidney function. The ratio was calculated by dividing the change from baseline B2M value by the urine creatinine value. B2M, beta 2 microglobulin (measured in mg/mmol).
Time Frame: Baseline, Week 96
Population: Safety Population. Some participants had withdrawn by Week 96.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 87 | 105
ratio | 0.542 [0.370 to 0.792] | 0.984 [0.684 to 1.416]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p < 0.0001, ANOVA — The model includes the following covariates: treatment, age, baseline biomarker value, baseline CD4, and gender; Estimates are calculated from an ANOVA model. Parameters are analyzed based on log transformed data

53. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in N-acetyl-B-glucosaminidase (NAG) as a Ratio to Urine Creatinine at Week 96
Description: Renal biomarkers were analyzed using urine samples collected from participants at baseline and Week 96. Renal biomarkers may be an indicator of various aspects of kidney function. The ratio was calculated by dividing the change from baseline NAG value by the urine creatinine value. NAG, N-acetyl-B-glucosaminidase (measured in micromoles per hour per millimole [umol/h/mmol]).
Time Frame: Baseline, Week 96
Population: as for outcome 51
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 103 | 120
ratio | 0.868 [0.774 to 0.974] | 0.939 [0.844 to 1.044]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.3323, ANOVA — The model includes the following covariates: treatment, age, and baseline biomarker value; Estimates are calculated from an ANOVA model. Parameters are analyzed based on log transformed data

54. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in Retinol Binding Protein (RBP) as a Ratio to Urine Creatinine at Week 96
Description: Renal biomarkers were analyzed using urine samples collected from participants at baseline and Week 96. Renal biomarkers may be an indicator of various aspects of kidney function. The ratio was calculated by dividing the change from baseline RBP value by the urine creatinine value. RBP, retinol binding protein (measured in micrograms per millimole [ug/mmol]).
Time Frame: Baseline, Week 96
Population: as for outcome 51
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 103 | 120
ratio | 1.099 [0.882 to 1.369] | 1.550 [1.247 to 1.927]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p < 0.0001, ANOVA — The model includes the following covariates: treatment, baseline biomarker value, baseline CD4, and gender; Estimates are calculated from an ANOVA model. Parameters are analyzed based on log transformed data

55. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in Procollagen Type 1 Amino-terminal Propeptide (P1NP) at Week 96
Description: P1NP is a bone biomarker that was analyzed using blood samples collected from participants at baseline and Week 96. Bone biomarkers may be an indicator of bone turnover.
Time Frame: Baseline, Week 96
Population: Safety Biomarker Population. Some participants had withdrawn by Week 96.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per Liter (ug/L)
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 94 | 114
micrograms per Liter (ug/L) | 1.2 [1.1 to 1.2] | 1.4 [1.3 to 1.5]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p < 0.0001, ANOVA — The model includes the following covariates: treatment, age, and baseline biomarker value; Estimates are calculated from ana ANOVA model. Parameters are analyzed based on log transformed data

56. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in Type 1 Collagen Cross-linked C-telopeptide at Week 96
Description: Bone biomarkers were analyzed using blood samples collected from participants at baseline and Week 96. Bone biomarkers may be an indicator of bone turnover.
Time Frame: Baseline, Week 96
Population: Safety Biomarker Population. Some participants had withdrawn by Week 96.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per Liter (ng/L)
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 94 | 114
nanograms per Liter (ng/L) | 89.9 [25.1 to 154.7] | 203.6 [143.3 to 264.0]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.0019, ANOVA — The model includes the following covariates: treatment, baseline biomarker value, and gender; Estimates are calculated from an ANOVA model

57. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in Osteocalcin at Week 96
Description: as for outcome 56
Time Frame: Baseline, Week 96
Population: Safety Biomarker Population. Some participants had withdrawn by Week 96.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/L
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 94 | 114
ug/L | 3.01 [0.87 to 5.14] | 5.79 [3.68 to 7.90]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.0019, ANOVA — The model includes the following covariates: treatment, age, baseline biomarker value, and baseline CD4; Estimates are calculated from an ANOVA model

58. Other Pre Specified Outcome: Exploratory Analysis of Change From Baseline in Bone Specific Alkaline Phosphatase (BSAP) at Week 96
Description: as for outcome 56
Time Frame: Baseline, Week 96
Population: Safety Biomarker Population. Some participants had withdrawn by Week 96.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/L
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Number analyzed (Participants) | 93 | 114
ug/L | 1.111 [-0.426 to 2.649] | 2.542 [1.028 to 4.056]
Statistical Analysis 1: Comparison: ABC/3TC FDC vs TDF/FTC FDC; Test type: Superiority or Other; p = 0.0266, ANOVA — The model includes the following covariates: treatment, baseline biomarker value, and baseline CD4; Estimates are calculated from an ANOVA model

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and adverse events (AEs) were collected in the Safety Population, comprised of all randomized participants who received at least one dose of study medication.
Arm/Group | ABC/3TC FDC | TDF/FTC FDC
Serious Adverse Events (participants affected / at risk) | 31/192 | 20/193
Other Adverse Events (participants affected / at risk) | 172/192 | 175/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABC/3TC FDC (N=192) | TDF/FTC FDC (N=193)
Drug hypersensitivity (Immune system disorders) | 5 | 1
Pneumonia (Infections and infestations) | 5 | 1
Hypersensitivity (Immune system disorders) | 3 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Immune reconstitution syndrome (Immune system disorders) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Eye infection toxoplasmal (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 1
Apathy (Psychiatric disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Porphyria non-acute (Congenital, familial and genetic disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABC/3TC FDC (N=192) | TDF/FTC FDC (N=193)
Nasopharyngitis (Infections and infestations) | 39 | 36
Influenza (Infections and infestations) | 12 | 14
Dizziness (Nervous system disorders) | 48 | 48
Headache (Nervous system disorders) | 17 | 29
Abnormal dreams (Psychiatric disorders) | 23 | 22
Insomnia (Psychiatric disorders) | 21 | 18
Sleep disorder (Psychiatric disorders) | 14 | 16
Depression (Psychiatric disorders) | 14 | 15
Diarrhoea (Gastrointestinal disorders) | 36 | 27
Nausea (Gastrointestinal disorders) | 17 | 16
Vomiting (Gastrointestinal disorders) | 12 | 11
Rash (Skin and subcutaneous tissue disorders) | 18 | 20
Fatigue (General disorders) | 14 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Bone density decreased (Investigations) | 5 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.